CLINICAL TRIAL: NCT01466309
Title: The Efficacy of Adjustable Thermoplastic Oral Appliances in Thai Patient With OSA
Brief Title: Efficacy of Adjustable Thermoplastic Oral Appliances in Patient With OSA
Acronym: ThaiSomnoguard
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Somnoguard in Thai OSA
Record Dates: First submitted 2011-11-01; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: OSA; Complication
Keywords: AHI; ESS; VAS; FOSQ; SF-36

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): patients treated with Somnoguard
  Interventions: Device: Somnoguard oral appliances

INTERVENTIONS:
Device: Somnoguard oral appliances — wearing somnogaurd daily at bedtime

SUMMARY:
Somnoguard, a titratable-thermoplastic oral appliances for the treatment of OSA, has been reported its safety and efficacy in Caucasians at least in the short-term. However, there has been no reports in Thai patients. The objectives of this study is to investigate its efficacy and safety in Thai patients with OSA.

DETAILED DESCRIPTION:
Fifty patients with any severity of OSA will be recruited according to the indications for oral appliance therapy in the practice parameters of the American Academy of Sleep Medicine (AASM)2006.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years with OSA
* AHI > 5
* Refused CPAP therapy

Exclusion Criteria:

* Poor oral hygiene
* Untreated TMD
* Inadequate healthy teeth (< 6)
* Severe or unstable medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea index | 1 year

SECONDARY OUTCOMES:
Number of Participants with Adverse Events" | 1 year
  Number of Participants with Adverse Events"

CONTACTS AND LOCATIONS:
Overall Officials: wish banhiran, MD, Principal Investigator — Yes
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand